CLINICAL TRIAL: NCT07152301
Title: Inflammatory Activation, Epigenetic Signature and Morpho-structural Alteration in a Cohort of Patients With Chronic Heart Failure and Permanent Non-valvular Atrial Fibrillation: a Cross-sectional Study
Brief Title: Inflammation, Epigenetics in CHF Patients With AF
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonino Tuttolomondo, Prof., University of Palermo
Other Study IDs: UPalermo8
Record Dates: First submitted 2025-08-16; First posted 2025-09-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Congestive Heart Failure Chronic; Atrial Fibrillation (Permanent)
Keywords: atrial fibrillation; congestive hearth failure; cytokine; miRNA
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma sample for evaluation of blood levels of cytokines and miRNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CHF and atrial fibrillation (CHF + AF): patients with chronic heart failure (CHF) and permanent non-valvular atrial fibrillation (AF)
- Patients with CHF and no atrial fibrillation (CHF no-AF): patients with CHF no prior history of atrial fibrillation

SUMMARY:
the goal of this case-control cross-sectional study is assessing in a cohort of patients with CHF and permanent AF

* The serum levels of some candidate cytokine variables and their relationship with some selected metabolic variables and some echocardiographic variables.
* the expression degree of some selected miRNA with a pathogenetic relation to atrial fibrillation and the related cardiac remodelling.
* to analyze the correlation between selected miRNA and the selected cytokines.

ELIGIBILITY:
Inclusion Criteria

* ≥18 years
* Left ventricular ejection fraction >40%
* New York Heart Association class II-IV symptoms
* NT-proBNP ≥600 pg/mL, or ≥900 pg/mL if AF was present on baseline electrocardiography

Exclusion Criteria

- Other AF subtypes (paroxysmal, persistent, long-standing persistent)

At least one of the following criteria:

* Acute heart failure
* NYHA IV
* NT-proBNP >4000 pg/mL
* Significant valvular disease
* Mechanical prosthesis
* Cardiovascular implantable devices
* Active malignancy
* Inflammatory or infectious diseases
* Severe renal (eGFR <30 mL/min/m²) or hepatic failure
* Chronic steroid/anti-inflammatory therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with chronic heart failure (CHF) and permanent non-valvular atrial fibrillation (AF), and consecutive patients with CHF, the same risk factors, but sinus rhythm and no prior AF history, admitted to the Internal Medicine and Stroke Care Ward of the "P. Giaccone" Hospital, Palermo
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
inflammation and structural cardiac remodelling | From January 2020 to May 2022
  in both arms of the study (AF + CHF and CHF no AF) a blood sample will be performed for the determination of serum values of inflammatory cytokines (CRP in mg/l; IL6 in pg/ml) and a transthoracic echocardiogram for the evaluation of the left atrial volume index in ml/m2 and the left atrial strain %

SECONDARY OUTCOMES:
epigenetic alterations and cardiac remodelling | From January 2020 to May 2022
  in both arms of the study (AF + CHF and CHF no AF) a blood sample will be performed for the determination of the expression degree of some selected miRNA with a pathogenetic relation to atrial fibrillation (hsa-miR-1-3p, hsa-miR-26a-5p, hsa-miR-21-5p in nmol/l), and a transthoracic echocardiogram for the evaluation of the left atrial volume index in ml/m2 and the left atrial strain %
inflammation and epigenetic alterations | From January 2020 to May 2022
  in both arms of the study (AF + CHF and CHF no AF) a blood sample will be performed for the determination of the expression degree of some selected miRNA with a pathogenetic relation to atrial fibrillation (hsa-miR-1-3p, hsa-miR-26a-5p, hsa-miR-21-5p in nmol/l), and a blood sample for the determination of serum values of inflammatory cytokines (CRP in mg/l; IL6 in pg/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine and Stroke Care Ward, Policlinic Hospital of Palermo, Sicily, Palermo, PA, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: August 2025-August 2030
Access Criteria: Professor Tuttolomondo will be responsible for responding to any queries regarding the protocol or results from those who request clarification via his institutional email address.

REFERENCES:
- [Background] Hage C, Michaelsson E, Linde C, Donal E, Daubert JC, Gan LM, Lund LH. Inflammatory Biomarkers Predict Heart Failure Severity and Prognosis in Patients With Heart Failure With Preserved Ejection Fraction: A Holistic Proteomic Approach. Circ Cardiovasc Genet. 2017 Feb;10(1):e001633. doi: 10.1161/CIRCGENETICS.116.001633. PMID 28100627
- [Background] Harada M, Van Wagoner DR, Nattel S. Role of inflammation in atrial fibrillation pathophysiology and management. Circ J. 2015;79(3):495-502. doi: 10.1253/circj.CJ-15-0138. Epub 2015 Feb 16. PMID 25746525
- [Background] Carr JJ, Hendel RC, White RD, Patel MR, Wolk MJ, Bettmann MA, Douglas P, Rybicki FJ, Kramer CM, Woodard PK, Shaw LJ, Yucel EK; American College of Cardiology Foundation; American College of Cardiology Foundation. 2013 appropriate utilization of cardiovascular imaging: a methodology for the development of joint criteria for the appropriate utilization of cardiovascular imaging by the American College of Cardiology Foundation and American College of Radiology. J Am Coll Radiol. 2013 Jun;10(6):456-63. doi: 10.1016/j.jacr.2013.03.019. Epub 2013 Apr 15. PMID 23598154